CLINICAL TRIAL: NCT00771082
Title: Osteoarthritis and Body Composition: Evaluation of Systematic Mediators
Status: Terminated | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Shari Ling, MD, National Institute on Aging
Other Study IDs: AG0109
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Knee Osteoarthritis
Keywords: inflammatory markers; bone markers; OA
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Banked serum and urine samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine the relationship between body composition and knee osteoarthritis, and effects of inflammatory, metabolic, and hormonal factors.

DETAILED DESCRIPTION:
Banked serum and urine specimens obtained from NIA Baltimore Longitudinal Study on Aging (BLSA) participants with and without knee OA will be used to determine inflammatory, metabolic, bone and joint biomarkers in an observational, case-control study. This study will be limited to BLSA data and samples that have already been acquired and stored.

The specific aims of this study are to:

1. Examine the association between prevalent radiographic osteoarthritis (OA), concurrently obtained inflammatory and metabolic mediator levels and change in bone density and bone markers over time subsequent to radiographic classification.
2. Determine levels of inflammatory, metabolic and bone markers, and body composition when radiographic OA was absent, and examine their relationship to the development of radiographic knee OA.

Adjustments will be made for age, gender, body mass index and level of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the BLSA who have had 1 or more DXA scans AND who were either classified as having radiographic knee OA (Kellgren & Lawrence 2 or higher) or as having no radiographic knee OA on two or more xrays (KL 0-1)

Exclusion Criteria:

* Diagnosis of rheumatoid arthritis
* Diagnosis of malignancy
* Reported use of prednisone and other immunosuppressive medications or insulin

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Baltimore Longitudinal Study on Aging
Sampling Method: Non-Probability Sample
Enrollment: 1033 (Actual)
Dates: Start 2003-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Changes in inflammatory marker c-reactive protein | 3 to 5 years

SECONDARY OUTCOMES:
Changes in other biomarkers: inflammatory, metabolic, bone, and joint | 3 to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Shari Ling, MD, Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute on Aging, Baltimore, Maryland, United States

REFERENCES:
- [Background] Felson DT, Zhang Y. An update on the epidemiology of knee and hip osteoarthritis with a view to prevention. Arthritis Rheum. 1998 Aug;41(8):1343-55. doi: 10.1002/1529-0131(199808)41:83.0.CO;2-9. No abstract available. PMID 9704632
- [Background] Hochberg MC, Lethbridge-Cejku M, Scott WW Jr, Reichle R, Plato CC, Tobin JD. The association of body weight, body fatness and body fat distribution with osteoarthritis of the knee: data from the Baltimore Longitudinal Study of Aging. J Rheumatol. 1995 Mar;22(3):488-93. PMID 7783067
- [Background] Lethbridge-Cejku M, Tobin JD, Scott WW Jr, Reichle R, Roy TA, Plato CC, Hochberg MC. Axial and hip bone mineral density and radiographic changes of osteoarthritis of the knee: data from the Baltimore Longitudinal Study of Aging. J Rheumatol. 1996 Nov;23(11):1943-7. PMID 8923372
- [Background] Sharif M, Shepstone L, Elson CJ, Dieppe PA, Kirwan JR. Increased serum C reactive protein may reflect events that precede radiographic progression in osteoarthritis of the knee. Ann Rheum Dis. 2000 Jan;59(1):71-4. doi: 10.1136/ard.59.1.71. PMID 10627432